CLINICAL TRIAL: NCT06825858
Title: A Phase I, Open-label, Multicenter, Dose-Escalating Study to Evaluate the Safety and Tolerability of KH658 Gene Therapy in Participants With Neovascular Age-related Macular Degeneration
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Origen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAN-2401
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KH658 Dose 1 (Experimental): KH658 One-Time Suprachroidal Space delivery Dose Level 1
  Interventions: Drug: KH658
- KH658 Dose 2 (Experimental): KH658 One-Time Suprachroidal Space delivery Dose Level 2
  Interventions: Drug: KH658
- KH658 Dose 3 (Experimental): KH658 One-Time Suprachroidal Space delivery Dose Level 3
  Interventions: Drug: KH658

INTERVENTIONS:
Drug: KH658 — KH658: AAV vector containing a coding sequence for an anti-VEGF protein

SUMMARY:
VAN-2401 is Phase I clinical trial to assess the safety and tolerability of KH658 in subjects with neovascular AMD. KH658 is gene therapy designed to deliver a protein which targets and blocks VEGF via an adeno-associated viral vector. The standard of care for patients with neovascular AMD are anti-VEGF treaments, which have demonstrated improvement in vision and reduction in fluid. A one time placement of a product which inhibits VEGF has the potential to reduce the patient burden of regular ocular injections.

ELIGIBILITY:
Inclusion Criteria:

-

1. Males and Females ages 50 to 85 (inclusive) with a study eye which meets the following criteria:

a. Previously received IVT treatment of anti-VEGF for neovascular AMD, with documented response to anti-VEGF therapy during the first 2 weeks of screening b. active macular CNV lesion secondary to AMD evidenced by SD-OCT c. Have a ETDRS BCVA letter score of 63 to 25 in the study eye at Screening for the first subject in each cohort (sentinel subject), followed by ETDRS BCVA letter score of 73 to 25 for the rest of the subjects each cohort; d. Are willing and able to sign the study written informed consent form (ICF).

Exclusion Criteria:

-

1. Have had any prior ocular or systemic treatment (investigational or approved) or surgery for the treatment of neovascular AMD except IVT anti-VEGF 2. Retinal pigment epithelial tears or rips at screening 3. Any history or presence of vitreous hemorrhage; 4. Have any condition preventing visual acuity improvement; 5. Have any other cause of CNV; prior pars plana vitrectomy or scleral buckling or retinal detachment surgery; macular hole, Epiretinal membrane or vitreo-macular traction; full thickness macular hole; 6. History of intraocular or periocular surgery in the prior 3 months; 7. Prior trabeculectomy or other filtration surgery (SLT or MIGS are permitted); 8. corneal transplant; 9. Any use of long-acting intraocular steroids, including implants, within six months prior; 10. Uncontrolled glaucoma; 11. Intraocular implant 12. Participated as a subject in any interventional clinical trial within 1 month prior; 13. Have received any gene or cell therapy product at any time in the past (either eye or systemically); 14. Have active intraocular inflammation in either eye at Screening or a history of uveitis in either eye 15.Have active ocular or periocular infection in either eye; 16. Have presence or history of scleromalacia in either eye;

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety | 52 Weeks
  type, severity and incidence of ocular and systemic AEs and SAEs
Safety | 52 Weeks
  Change in Best Corrected Visual Acuity
Safety | 24Weeks
  type, severity and incidence of ocular and systemic AEs and SAEs
Rescue Injections | 24Weeks
  Mean Number of Rescue Injections
Rescue Injections | 52Weeks
  Mean Number of Rescue Injections

SECONDARY OUTCOMES:
Safety | 24 Weeks
  Change in Best Corrected Visual Acuity

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Kanghong Investigative Site, Phoenix, Arizona
  - Kanghong Investigative Site, Lemont, Illinois
  - Kanghong Investigative Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No